CLINICAL TRIAL: NCT04197518
Title: Evaluation the Neurocognitive Functions Among Children With Enlargement Adenoid and Tonsils, Before and After Tonsillectomy or Adenotonsillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0042-18-HYMC
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Child Neurocognitive Function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children With Enlargement Adenoid and Tonsils (Experimental): Children With Enlargement Adenoid and Tonsils
  Interventions: Diagnostic Test: neuro trax system and a neurology test.

INTERVENTIONS:
Diagnostic Test: neuro trax system and a neurology test. — the neurology will check the patience before and after tonsillectomy or adenotonsillectomy usung the neurotrax system, these parameters will be measured in this system : Non verbal memory, Go no go test, stroop interference, Visual spatial processing, Staged information processing speed, "catch" game, problem solving.

SUMMARY:
Evaluation the Neurocognitive Functions Among Children With Enlargement Adenoid and Tonsils, Before and After Tonsillectomy or Adenotonsillectomy

ELIGIBILITY:
Inclusion Criteria:

* children between 6-18 years old.
* children with enlarged tonsils or adenoids.
* a sleep lab test before the procedure.

Exclusion Criteria:

* children under 6 years old and above 18 years old.
* patience that treated in ADHD / ADDOR with other neurocognitive disorder.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Functions Among Children | 2 years
  neurology test using neuro trax system , to evaluate Neurocognitive Functions Among Children With Enlargement Adenoid and Tonsils, Before and After Tonsillectomy or Adenotonsillectomy